CLINICAL TRIAL: NCT00721357
Title: Skeletal Muscle Properties and the Metabolic Cost of Walking Post-Stroke
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: B6341-W
Record Dates: First submitted 2008-07-21; First posted 2008-07-24 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2018-12

CONDITIONS: Stroke
Keywords: muscles; work; Magnetic Resonance Imaging; control groups
MeSH Terms: conditions — Stroke | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — None retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stroke: Stroke subjects
  Interventions: Behavioral: Treadmill walking; Other: Magnetic resonance spectroscopy
- Control: neurologically healthy subjects
  Interventions: Behavioral: Treadmill walking; Other: Magnetic resonance spectroscopy

INTERVENTIONS:
Behavioral: Treadmill walking — Subjects will perform treadmill walking at a self-selected velocity
Other: Magnetic resonance spectroscopy — Muscle oxidative capacity will be assessed via Magnetic resonance spectroscopy (31P-MRS)

SUMMARY:
Of the ~700,000 persons who suffer a stroke each year, only 50% recover the ability to perform unlimited community walking. One mechanism contributing to locomotor dysfunction post-stroke is an increased metabolic cost of walking relative to neurologically healthy individuals 2-4. This increased cost likely limits the amount of walking performed, which further reduces functional capacity, thus contributing to long-term spiral of disability and decreased quality of life in these persons. In addition to increased metabolic cost, increased estimates of mechanical work are also characteristic of hemiparetic walking 2,29. Interestingly, although estimates of mechanical work reflect work done by locomotor muscles, little is known about the impact that peripheral muscle properties have on estimates of mechanical work. Furthermore, questions concerning how these properties relate to the increased metabolic cost of walking remain unanswered. The short-term objective and purpose of the proposed research is to determine the extent to which peripheral muscle characteristics, as well as estimates of muscle mechanical energy expenditure (MMEE), relate to the metabolic cost of walking post-stroke.

DETAILED DESCRIPTION:
A guiding principle of the proposed research is that skeletal muscle is the building block of all movement and, as such, muscle dysfunction can ultimately limit the gains possible from rehabilitation intervention. Therefore, maximal gains will be made only when central nervous system adaptations access peripheral muscle that is fully capable of supporting the increased activity.

The primary hypothesis is that in persons with hemiparesis following stroke, alterations in the metabolic properties of peripheral skeletal muscles, in combination with greater mechanical work, contribute to the increased metabolic cost of walking. A secondary hypothesis is that locomotor training induces adaptations in lower extremity skeletal muscle resulting in improved mechanical and metabolic efficiency. In order to test these hypotheses, the following three specific aims will be addressed:

Aim 1: Determine the in-vivo metabolic characteristics of the ankle plantar flexor muscles in persons with chronic post-stroke hemiparesis and neurologically healthy individuals. In-vivo muscle metabolic properties will be assessed via phosphorous magnetic resonance spectroscopy (31P-MRS). Specifically, we will measure the resting phosphorylation potential as well as the in-vivo oxidative capacity of the ankle plantar flexor muscles. We hypothesize that individuals with chronic hemiparesis will exhibit reductions in oxidative capacity as well as an increased resting phosphorylation potential relative to age-, gender-, height- and weight-matched control subjects. We suggest these adaptations, which are characteristic of a less energetically efficient muscle, contribute to an increased metabolic cost beyond that resulting from potential increases in mechanical work performed by locomotor muscles.

Aim 2: Quantify metabolic cost as well as muscle mechanical energy expenditure during walking in persons with chronic post-stroke hemiparesis and neurologically healthy individuals. Post-stroke hemiparesis is associated with a variety of motor control problems that include abnormal synergistic organization of movement as well as altered temporal sequencing of muscle activity 5,10,11. Since muscle excitation during normal walking is believed to be very efficient 8,9,33 it is likely that altered muscle coordination post-stroke, reflected in increased mechanical work, is one factor contributing to the increased metabolic cost of walking. We hypothesize that the metabolic cost of walking post-stroke will be elevated relative to controls at matched speeds. Additionally, a measure of mechanical work, muscle mechanical energy expenditure (MMEE), will be elevated post-stroke, reflective of mechanically inefficient movement strategies and causal to a portion of the increased metabolic cost of walking.

Aim 3: Determine the impact of 12 weeks of locomotor training on in-vivo muscle metabolic properties, the metabolic cost of walking as well as MMEE in persons with chronic post-stroke hemiparesis. There is emerging evidence that chronic neurologic deficits due to stroke can be improved through intensive, repetitive task-oriented motor training (e.g. locomotor training). The basis for locomotor training (LT) improvements is thought to involve mechanisms of central neuroplasticity that are responsive to fundamental principles of motor learning 37,38,39. In addition, our pilot data demonstrate that LT may also result in peripheral adaptations in the plantar flexor muscles. Thus, the potential seemingly exists to induce both central and peripheral adaptations with this intervention strategy. We expect that LT will attenuate existing deficits, resulting in an increased oxidative capacity and a decreased resting phosphorylation potential in ankle plantar flexor muscles. In addition, LT will result in a reduced MMEE and a reduced metabolic cost of walking, reflective of improved mechanical and metabolic efficiency. We believe it will prove important to describe adaptations in walking mechanics as well as within peripheral muscle that occur following LT and relate them to the metabolic cost of walking. In addition, continued deficits will reflect a need for additional or adjunctive intervention strategies, thus providing information on how to modify or augment future rehabilitation interventions in order to improve individual outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80;
* stroke within past 6 months - 5 years;
* residual paresis in the lower extremity (LE) (Fugl-Meyer motor score <34);
* ability to sit unsupported for 30 sec;
* ability to walk at least 10 ft with maximum 1 person assist;
* self selected 10 meter gait speed < 0.8 m/s; and
* provision of informed consent.

Exclusion Criteria:

* Unable to ambulate at least 150 feet prior to stroke, or experienced intermittent claudication while walking < 200 meters;
* history of congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living;
* History of chronic obstructive pulmonary disease or oxygen dependence;
* Preexisting neurological disorders, dementia or previous stroke;
* History of major head trauma;
* Legal blindness or severe visual impairment;
* history of significant psychiatric illness;
* Life expectancy <1 yr;
* Severe arthritis or orthopedic problems that limit passive range of motion (ROM);
* post-stroke depression (PHQ-9 10);
* History of deep vein thrombosis (DVT) or pulmonary embolism within 6 months;
* Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions;
* Severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest;
* Previous or current enrollment in a clinical trial to enhance motor recovery;
* Presence of non-magnetic resonance (MR) compatible implants or devices, pregnancy or severe claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris M. Gregory, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stroke: those with condition
  Treadmill walking: Subjects will perform treadmill walking at a self-selected velocity
  Magnetic resonance spectroscopy: Muscle oxidative capacity will be assessed via Magnetic resonance spectroscopy (31P-MRS)
- Control: those without condition
  Treadmill walking: Subjects will perform treadmill walking at a self-selected velocity
  Magnetic resonance spectroscopy: Muscle oxidative capacity will be assessed via Magnetic resonance spectroscopy (31P-MRS)
Period: Overall Study
Arm/Group | Stroke | Control
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stroke | Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (9.2) | 54.2 (5.1) | 57.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 8 | 10 | 18
walking speed [Mean (Standard Deviation); unit: meters per second] — The overground speed the individuals walk when instructed to "walk at you normal comfortable speed".
  meters per second | 0.57 (0.23) | 1.17 (0.15) | 0.87 (0.20)
muscle oxidative capacity [Mean (Standard Deviation); unit: millimolar inorganic phosphate] — This measures specific compounds in leg muscles to estimate how well they would perform repeated physical tasks (e.g. walking).
  millimolar inorganic phosphate | 5.1 (0.87) | 3.2 (0.56) | 4.2 (0.72)
muscle mechanical energy expenditure [Mean (Standard Deviation); unit: Joules per kg] — This is a calculation of how much work is done by each joint (i.e. ankle, knee and hip) of each leag during walking.
  Joules per kg | 374 (161) | 242 (66) | 309 (112)

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Consumption During Walking
Description: Amount of oxygen consumed during walking at self-selected speed normalized to speed
Time Frame: within one week of enrollment
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Stroke | Control
Number analyzed (Participants) | 15 | 15
ml/kg/min | 11.25 (.76) | 4.46 (.27)

2. Secondary Outcome: Muscle Mechanical Energy Expenditure
Description: mechanical work done by lower extremity joints
Time Frame: one time measure within one week of enrollment
Population: Individuals following stroke and matched non-stroke individuals. Sample size differences reflect the inability of some subjects to walk on the instrumented treadmill at speeds necessary to collect the kinematic data.
Measure: Mean (Standard Deviation); unit: joules per kilogram meter
Arm/Group | Stroke | Control
Number analyzed (Participants) | 12 | 12
joules per kilogram meter | 5.66 (1.89) | 3.61 (1.42)

3. Secondary Outcome: Magnetic Resonance Spectroscopy of Muscle Metabolic Properties
Description: time constant indicating the time for recovery in muscle phosphocreatine levels following exercise as a metric of muscle oxidative capacity.
Time Frame: within one week of enrollment
Population: Sample size differences reflect the fact that some subjects are either incompatible with imaging procedures because they are either unable to lie still for the time necessary to collect these data, are claustrophobic or have metal somewhere in their body that prevents imaging.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Stroke | Control
Number analyzed (Participants) | 9 | 6
seconds | 43.22 (9.8) | 35.39 (8.26)

ADVERSE EVENTS:
Arm/Group | Stroke | Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stroke (N=15) | Control (N=15)
fall at home (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject reported a fall int he home but did not result in injury

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes